CLINICAL TRIAL: NCT03112824
Title: Functional Assessment of Ashwagandaha Root Extract During Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: #5170083
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Stress Reaction; Sleep Disturbance; Craving; Obesity
MeSH Terms: conditions — Fractures, Stress; Parasomnias; Obesity

STUDY DESIGN:
Intervention Model Description: If the PSS score is than 20, those patients who are interested in participating are consented to the Ashwagandha study. The patients will then be randomized in a double-blind fashion to receive a 31 day supply of study capsules which will be either Ashwagandha 300mg twice a day or identical placebo capsules in a 1:1 ratio. They will be given careful directions into the use of the study capsules and will be asked to mark a daily log (See addendum #3: Treatment Log) of taking the capsules in the morning and at night.
Who Masked: Participant, Care Provider, Investigator
Masking Description: A designated MD who is not involved in the study design, application, or interpretation will be available to unblind study participants when medically indicated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ashwagandaha Root Extract Capsule (Experimental): Participants will take one 300 mg. Ashwaganda capsule twice a day for 12 weeks.
  Interventions: Dietary Supplement: Ashwagandha Root Extract Capsule
- Placebo Capsule (Placebo Comparator): Participants will take one placebo capsule twice a day for 12 weeks.
  Interventions: Other: Placebo Capsule

INTERVENTIONS:
Dietary Supplement: Ashwagandha Root Extract Capsule — Participants will take one 300 mg capsule of Ashwagandaha Root Extract orally twice a day for 12 weeks.
  Arms: Ashwagandaha Root Extract Capsule
Other: Placebo Capsule — Participants will take one placebo capsule orally twice a day for 12 weeks.
  Arms: Placebo Capsule

SUMMARY:
Patients who are involved in a clinical protocol driven 12 week medical weight loss intervention will be randomized to receive either a placebo or 600 mg of an ashwagandha root extract. The study endpoints are primarily the patients self-reported perception of life stress and sleep quality. The working hypothesis of this study is that the addition of aschwagandha to .the medical weight loss program will improve the self-reported perception of life stress and sleep quality

DETAILED DESCRIPTION:
During this 12-week medical weight loss program, the randomized patients will also have a baseline measurements and final measurements of blood for selected adipokines , cytokines, and telomerase measurements

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. BMI of 27 kg/m2 with comorbidities or 30 kg/m2 and above
  2. Perceived Stress Scale (PSS) score of ≥ 20 at screening
  3. Age 18 to 70 years
  4. Generally healthy male or female in the judgement of the principal investigator.
  5. Able to attend the testing site at CHP.
  6. Access to a computer and are able to enter information into the computer

Exclusion Criteria:

* Exclusion criteria (Justification of exclusion group based on demographics or their vulnerability)

  1. Taking chronic anti-anxiety, anti-obesity (other than phentermine) or anti-insomnia medication on a regular basis and unwilling to stop taking these classes of medications for the duration of the 12 week trial.
  2. Adults unable to consent
  3. Individuals who are not yet adults (infants, children, teenagers)
  4. Pregnant women
  5. Prisoners
  6. Nursing an infant
  7. Currently undergoing cancer treatment
  8. Untreated hypertension, diabetes or cardiac arrhythmias
  9. Dieting to lose weight in the last month
  10. Started within the last 14 days or plan to start taking:
* Birth control pills
* Hormone supplements (Estrogen/Progesterone etc)
* MAO inhibitors, Oral Corticosteroids, Tricyclic antidepressants, SSRI's (except Fluoxetine),

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale PSS | 12 weeks
  Standardized questionnaire

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index PSQI | 12 weeks
  Standardized questionnaire
Food Craving Questionnaire - Trait FCQ-T | 12 weeks
  Standardized questionnaire
Three-Factor Eating Questionnaire TFEQ | 12 weeks
  Standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Warren R Peters, MD MPH, Principal Investigator — LLU Administrator
Locations (1):
- Loma Linda University Center for Health Promotion, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plans to share IPD